CLINICAL TRIAL: NCT00167466
Title: Randomized, Double-blind, Placebo-controlled Crossover Trial of the Soladey-3 Toothbrush on Periodontal Disease Indices in Patients With Mild-to-moderate Periodontal Disease
Brief Title: Placebo Controlled Trial of a Titanium Dioxide Semiconductor Toothbrush on Mild-to-moderate Gum Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: Shiken Corporation (Industry)
Responsible Party: Dr. Gerry Uswak, University of Saskatchewan
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Bio-REB 05-20
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2010-10-28 (Estimated); Status verified 2010-10

CONDITIONS: Periodontal Diseases
Keywords: periodontal disease; toothbrush; titanium dioxide semiconductor; mild-to-moderate periodontal disease; adult patients 18 to 70 years of age
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): 4 week brushing with experimental Soladey-3 toothbrush followed by 4 week washout period followed by 4 week brushing with placebo Soladey-3 toothbrush
  Interventions: Device: Soladey-3 toothbrush
- B (Placebo Comparator): subjects to brush with Placebo Soladey-3 toothbrush for 4 weeks followed by a 4 week washout followed by 4 week brushing with experimental Soladey-3 toothbrush
  Interventions: Device: Placebo Soladey-3 toothbrush

INTERVENTIONS:
Device: Soladey-3 toothbrush — subject to brush with experimental Soladey-3 brush for 4 week
  Arms: A
Device: Placebo Soladey-3 toothbrush — subjects will brush with placebo Soladey-3 toothbrush for 4 weeks
  Arms: B

SUMMARY:
The effects on indices of gingivitis/periodontitis will differ between study arms in which the titanium dioxide semiconductor toothbrush is used, compared to an otherwise identical toothbrush with an inert resin core in place of the titanium dioxide semiconductor.

DETAILED DESCRIPTION:
Organic acid producing anaerobic bacteria are implicated in the development and progression of gingivitis and periodontal disease (Brill, 1962; Kleinberg, 1974). The disease process manifests as periodontal inflammation and tissue destruction (Oliver et al, 1969). Although relatively crude methods are used for routine clinical diagnosis and monitoring of periodontal disease (eg, probing for gingival pocket depth and bleeding), sensitive and reproducible measures of periodontal disease have been validated (Oliver et al, 1969; Löe et al, 1965; Egelberg, 1964; Golub et al, 1976; Borden et al, 1977).

By the Lewis definition, an acid is an electron pair acceptor. In the presence of light &/or electrical induction, valence electrons from a wetted titanium dioxide (TiO2) semiconductor will donate electron pairs to neutralize organic acids. Whereas a tooth surface is negatively charged, plaque has a net positive charge, and in part, ionic attraction contributes to the adherence of plaque to the tooth surface. Donating electrons to the plaque will alter polarity and diminish the ionic attraction between the plaque and the tooth surface (iontophoretic effect).

Thus, in addition to the established mechanical benefits of brushing, the flow of electron pairs for disrupting ionic bonding of plaque to the tooth surface and neutralizing bacterial organic acids, may confer an advantage over a conventional toothbrush (Hoover et al, 1992; Niwa et al, 1989; Kusunoki et al, 1986). There is some evidence that the electrons may also interact with bacterial coenzyme-A to have an antibacterial effect (Morioka et al, 1988; Onoda et al, 1996).

ELIGIBILITY:
Inclusion Criteria:

* 30 to 70 yrs of age
* mild-to-moderate periodontal disease
* dentulous

Exclusion Criteria:

* any unstable medical condition
* pocket depth > 5 mm

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2005-10; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
gingivitis index | 4 measurements 4 weeks apart
plaque index | 4 measurements 4 weeks apart

SECONDARY OUTCOMES:
subjective comments re: functionality of of the Soladey-3 toothbrush compared to conventional toothbrush. | End of study assessment

CONTACTS AND LOCATIONS:
Overall Officials: Gerry Uswak, Principal Investigator — University of Saskatchewan
Locations (1):
- University of Saskatchewan College of Dentistry, Saskatoon, Saskatchewan, Canada